CLINICAL TRIAL: NCT01183351
Title: Pilot Study of a Multidisciplinary Intervention for Challenging Behaviour (Agitation) in Patients With Dementia
Brief Title: Multidisciplinary Intervention for Challenging Behaviour (Agitation) in Patients With Dementia
Acronym: TID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Norwegian Medical Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MID
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2011-05

CONDITIONS: Dementia
Keywords: Dementia; Agitation; Challenging behaviour; Behavioural and psychological symptoms in dementia (BPSD)
MeSH Terms: conditions — Dementia; Psychomotor Agitation | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychosocial intervention (Experimental): This is a single-group pilot-study
  Interventions: Behavioral: Psychosocial intervention

INTERVENTIONS:
Behavioral: Psychosocial intervention — Multidisciplinary Intervention for challenging behavior in patients with Dementia (MID) is developed in clinical practice in nursing homes as an answer to the need of a systematic and simple tool for the nursing home health workers to meet agitation. The model is based on the theoretical framework of cognitive behavioural therapy (CBT) where human behaviour is understood as always acting under the influence of biological, social and psychological factors. The systematic and structured approach of CBT to problem solving is central and is transformed in the model to meet the specific characteristics of challenging behaviour in dementia.
  Other Names: Multidisclinary Intervention in Dementia patients; Psychosocial intervention for challenging behavior

SUMMARY:
The increasing prevalence of dementia is a major challenge to the health authorities in most countries. Nearly all the persons suffering from dementia experience behavioural and psychological symptoms (BPSD). The prevalence of BPSD is particularly high in nursing homes. BPSD are often treated with psychotropic drugs even though the evidence for effect is minimal and the risk of serious adverse events is considerable. All the major treatment recommendations advise that non-pharmacological measures should be applied first when treating BPSD even though the evidence for such treatment is limited. The investigators will conduct a pilot study of a non-pharmacological treatment for BPSD. The method has been developed in Norway and has already been implemented in a number of nursing homes in the county of Nordland.

DETAILED DESCRIPTION:
Intervention description:

Initially the intervention group will receive education about dementia, BPSD, quality of care and use of psychotropic drugs Subsequently, staff in the nursing home will receive training in the intervention method: MID. Two or three nurses from each nursing home will receive more intensive training in the method to ensure effective implementation of the method in daily practice. After this initial period that will last for four weeks, trained research nurses will visit each nursing home every fortnight ensuring that the intervention is properly implemented and thereby assure adherence to the treatment protocol.

Description of the intervention Multidisciplinary Intervention model for challenging behaviour in Dementia, MID, consists of three stages: a registration-observation stage, a staff guiding stage, and an evaluation stage.

1. Registration-observation stage:

   The nurses use a daily registration sheet for the actual types of behaviour that are challenging. This ensures that the behaviour is properly observed on a daily basis.

   The next step in the registration-observation stage is:
   * Collection of the medical history by the nursing home nurses
   * Standard physical examination by the nursing home physician
   * Critical review of medication by the nursing home physician
   * Pain assessment (clinical), by the nursing home physician
   * Assessment of the type and degree of dementia by the nursing home physician
   * Assembly of the patients personal history by the nursing homes nurses After completion of the registration-observation stage (lasting 1 day up to 4 weeks) the staff guiding stage starts.
2. Staff guiding stage - guiding meeting The trained nurses from the nursing home set a meeting for 1-1,5 hours for the nursing home health workers. The meeting is lead by the nursing home nurses and the nursing home physician.

   The meeting follows a structured agenda and is conducted following the principles of problem solving in cognitive behavioural therapy taking into account one type of challenging behaviour at a time. Results from the registration-observation stage are presented at the beginning of the meeting. (A 5-column sheet, based on classical cognitive change thoughts records, is used to structure problem solving during the meeting: 1.facts, 2.interpretations (thoughts), 3.feelings, 4. solutions/actions and 5. evaluation)
3. Evaluation stage This stage starts just after the guiding meeting and is conducted by the nursing home nurses. The nurses continue the same registration of the behaviour on a daily basis as in the registration-observation stage for the next 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for inclusion if they have a possible or probable dementia diagnosis and clinically significant agitation score 6 or higher (as measured by the CMAI: Cohen-Mansfield Agitation Behaviour
* A permanent stay in nursing home of at least 4 weeks
* Given verbal or written assent for participation or has written consent given on their behalf by their next of kin

Exclusion Criteria:

* Lack of consent, terminal state,unremitting pain.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Agitation measured by the C-MAI (The Cohen-Mansfield Agitation Inventory) | 8 months

SECONDARY OUTCOMES:
The Cornell scale for depression in dementia (CSDD) | 8 months
Neuropsychiatric Inventory (NPI ) which measures neuropsychiatric symptoms and behaviour | 8 months
Lawton's self-maintenance scale (Lawton and Brody 1969), which measures function in activities of daily living (ADL) | 8 months
Quality of life in Alzheimers's Disease (QUALID) (Weiner et al. 2000), which measures quality of life | 8 months
Staff measures: Psychosocial factors in work life will be measured by a scale developed by Sund (1992). | 8 months
Use of antipsychotic drugs | 8 months
Staff measures:P-cat:Person-centered Care Assessment Tool | 8 months
  Measure of the degree of person-centered dementia care in the unit

CONTACTS AND LOCATIONS:
Overall Officials: Geir Selbaek, MD PhD, Study Chair — Sykehuset Innlandet HF
Locations (1):
- Department for Research and Development, Innlandet Hospital Trust, Hamar, Norway